CLINICAL TRIAL: NCT02476929
Title: AssEssment and New Perspectives on Pathophysiogenesis, detectiOn and Use of NAsal Nitrous Oxide and the Electronic Nose (EPONA Project)
Brief Title: Detection and Use of Nasal Nitrous Oxide and the Electronic Nose
Acronym: EPONA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Universitat Autonoma de Barcelona (Other); Sociedad Española de Alergología e Inmunología Clínica (Unknown); Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IIBSP-ONA-2011-146
Record Dates: First submitted 2015-03-02; First posted 2015-06-22 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Allergic Rhinitis; Non-Allergic Rhinitis; Nasal Polyps
Keywords: Electronic nose; Nasal nitrous oxide; Allergic Rhinitis; Non-Allergic Rhinitis; Nasal polyps
MeSH Terms: conditions — Rhinitis, Allergic; Common Cold; Nasal Polyps | interventions — Electronic Nose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nasal nitrous oxide (Active Comparator): Mesurement of Nasal nitrous oxide in all groups: allergic rhinitis, non-allergic rhinitis, nasosinusal polyps and healthy group
  Interventions: Device: Nasal nitrous oxide
- Electronic nose (Active Comparator): Measurement with the Electronic nose in all groups: allergic rhinitis, non-allergic rhinitis, nasosinusal polyps and healthy group.
  Interventions: Device: Electronic nose

INTERVENTIONS:
Device: Nasal nitrous oxide — Electrochemical device (NOVario Analizer FILT), to determine reference values of Nasal nitrous oxide.
  Arms: Nasal nitrous oxide
Device: Electronic nose — To determine reference values of different patterns of specific volatile organic compounds with the electronic nose (Cyranose 320®).
  Arms: Electronic nose

SUMMARY:
Introduction: Rhinitis, sinonasal polyposis (SP) and asthma are diseases whose pathogenesis is based on inflammation. This will determine the presence of disease, its evolution and its treatment. It is therefore very important to develop and validate methodologies that allow us to noninvasively detect inflammation of the airways. Thus, just as exhaled nitric oxide (FeNO) has been studied as an important non-invasive marker of inflammation of the lower airways, nasal nitric oxide (nNO) may be a good marker of nasal inflammation. Furthermore, the electronic nose is an electronic nanosensor device capable of detecting specific volatile organic compounds (VOCs) that can be used as a non-invasive biomarker of biochemical processes in different diseases whose pathophysiology is also based on inflammation.

Objective: To determine reference values of nNO and different patterns of VOCs in healthy individuals, individuals with allergic rhinitis (AR) and non-allergic rhinitis and individuals with SP and asthma.

Methodology: Prospective, controlled study. Four groups will be included: Healthy subjects, patients with AR, non-allergic rhinitis and patients with SP and asthma (n=252). Prick-test to pneumoallergens will be performed. Determination of FeNO, nNO, lung function tests, measurement of VOCs by the electronic nose and blood samples will be taken. Bilateral nasal endoscopy and sample collection using the technique of brushing of mucosa and the placement of filter papers, for the study of nasal cytology and mediators of inflammation.

DETAILED DESCRIPTION:
Assessment of nasal and bronchial inflammation:

Rhinitis (allergic and non-allergic), SP and asthma are diseases that are characterized by processes whose pathogenesis is based on inflammation. Inflammation of the airways can be assessed directly or indirectly. The techniques for assessing inflammation directly can be divided into invasive techniques and non-invasive techniques.

Within invasive techniques we include those which require nasal or bronchial endoscopy such as biopsy. However, the applicability of these invasive methods has many limitations because they are not without risks and/or complications. They also require considerable experience to implement. It is therefore very important to develop and validate new methods that allow us to non-invasively detect inflammation of the upper and lower airways.

Nitrous oxide (NO): Is synthesized from the amino acid L-arginine by the action of the enzyme nitric oxide synthase (NOS). Three isoforms of this enzyme are known: nNOS or NOS1, which predominates in nervous tissue; iNOS, inducible NOS or NOS2, induced by an agent that activates the immune system; and eNOS, endothelial NOS or NOS3, constituent of the vascular endothelium. Since iNOS is found in different cells of the respiratory tract and is induced by various inflammatory cytokines, NO is considered to be an excellent marker for airway inflammation. Thus, just as exhaled nitric oxide (FeNO) is considered a good non-invasive marker of inflammation of the lower airways, nasal nitric oxide (nNO) potentially appears be a good marker of nasal inflammation.

Nasal nitric oxide (nNO): Some authors describe reference values for nNO up to one hundred times higher than those for FeNO. However, until now normal levels of nNO in different nasal diseases and in healthy individuals have not been established because the published results vary widely. Dotsch et al. in 1996 published a series of 67 healthy subjects in which they found mean nNO values in a healthy population of 96±47 ppb. A year later Ferguson studied 82 healthy patients and published mean normal values of nNO of 1197±361 ppb. Additional papers were published subsequently, but the results remained quite diverse.

As for the reference values in patients with rhinitis, data published so far are also contradictory. Some authors show that nNO is higher in patients diagnosed with rhinitis, especially in patients with AR. However, other studies have not observed differences in levels of nNO in patients diagnosed with rhinitis compared to the normal population.

The electronic nose: Is a new technique which is based on the detection of VOCs present in the gas phase of the human respiration and that can be detected by chromatography and mass spectrometry sensors. It consists of a device made up of several nanosensors that when exposed to volatile particles undergo specific changes in their electrical resistance, resulting in a pattern or profile of VOCs by logarithmic regression. These VOC patterns can be used as non-invasive biomarkers of several biochemical processes that occur in different diseases whose pathogenesis is based on inflammation. For example, in diseases of the airways they have been used successfully in comparing patterns of VOCs in patients with chronic obstructive pulmonary disease (COPD) and asthma. This technique's potential applicability in biomedicine is enormous.

In short, both measuring nNO and determining patterns of VOCs by the electronic nose are non-invasive methods that can help in the diagnosis and monitoring of certain respiratory diseases. However, in the case of nNO currently available studies show very different and conflicting results and in the case of the determination of VOCs by electronic nose there are very few papers published to date. It is therefore vital to design a study that allows us to clarify the potential utility of non-invasive markers of inflammation such as determination of nNO and determination of the different patterns of VOCs by electronic nose in healthy patients, in patients diagnosed with AR and non-allergic rhinitis and in patients with associated SP and asthma.

Working Hypothesis: Rhinitis, SP and asthma are prevalent diseases that cause considerable morbidity. Since the substrate of these diseases lies in inflammation, our group of investigators believe that the study of inflammation is one of the most interesting aspects for assessment and management of these diseases. Similarly to how measuring FeNO is being used as a good marker of bronchial inflammation, measuring nNO and determining patterns of VOCs by the electronic nose could also be two good non-invasive markers of upper and/or lower (in the case of VOCs) airway inflammation. However, although in recent years there have been some studies on the origin, function and utility of measuring nNO and the use of the electronic nose in respiratory disease, there are still many questions that remain in reference to these two techniques.

ELIGIBILITY:
Inclusion criteria:

Sample of healthy individuals: Non-atopic individuals will be considered when skin prick skin tests with a standard battery of pneumoallergens are negative.

* Individuals with nasal endoscopy not showing inflammatory lesions or anatomic abnormalities and who have an acoustic rhinometry compatible with normal values.
* No sign of any acute infectious process during the four weeks preceding the study.
* Signed informed consent.

Sample of individuals with Allergic Rhinitis: Atopic patients sensitized by skin prick testing and specific IgE determination to at least one perennial allergen.

* Patients with symptoms compatible with persistent moderate or severe AR as rated by the ARIA 2008 guide of at least two years of evolution.
* No acute infectious process during the four weeks preceding the study.
* Signed informed consent.

Sample of individuals with non-allergic rhinitis: The subject will be considered non-atopic when skin prick skin tests with a standard battery of pneumoallergens are negative.

* Patients with symptoms of sneezing, watery rhinorrhea, nasal itching and/or nasal obstruction of at least two years evolution.
* No acute infectious process during the four weeks preceding the study.
* Signed informed consent.

Sample of individuals diagnosed with Sinunasal Polyposis and asthma: Patients diagnosed with asthma by clinical and lung function tests.

* SP patients diagnosed by performing nasal endoscopy and CT of the paranasal sinuses.
* Could be non-atopic patients or present any concomitant allergic diseases.
* No acute infectious process during the four weeks preceding the study.
* Signed informed consent.

Exclusion criteria for all groups:

* Smoker with history of more than 10 pack-years.
* Pregnancy.
* Having been treated with nasal or systemic drugs that may alter nasal resistance (vasoconstrictors, anticholinergics, corticosteroids, antihistamines, immunosuppressants and/or immunomodulators) during the past three weeks.
* History of nasal surgery.
* Having an autoimmune or inflammatory systemic disease.
* Having an established diagnosis of intrinsic or extrinsic asthma (except polyposis group).
* Individuals with pathological nasal endoscopy.
* Suffering from a neoplastic disease.
* Having been treated with nasal or systemic drugs that may alter nasal resistance (vasoconstrictors, anticholinergics, corticosteroids, antihistamines, immunosuppressants and/or immunomodulators) during the past three weeks.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2013-01; Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Values of nNO measure as parts per billions (ppb) | 12 months
Values of the electronic nose measure as volatile organic compounts (VOCs) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lorena Soto-Retes, physician, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Lorena Soto-Retes, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dragonieri S, Schot R, Mertens BJ, Le Cessie S, Gauw SA, Spanevello A, Resta O, Willard NP, Vink TJ, Rabe KF, Bel EH, Sterk PJ. An electronic nose in the discrimination of patients with asthma and controls. J Allergy Clin Immunol. 2007 Oct;120(4):856-62. doi: 10.1016/j.jaci.2007.05.043. Epub 2007 Jul 20. PMID 17658592
- [Result] Silkoff PE, Robbins RA, Gaston B, Lundberg JO, Townley RG. Endogenous nitric oxide in allergic airway disease. J Allergy Clin Immunol. 2000 Mar;105(3):438-48. doi: 10.1067/mai.2000.104938. PMID 10719291
- [Result] Lundberg JO, Farkas-Szallasi T, Weitzberg E, Rinder J, Lidholm J, Anggaard A, Hokfelt T, Lundberg JM, Alving K. High nitric oxide production in human paranasal sinuses. Nat Med. 1995 Apr;1(4):370-3. doi: 10.1038/nm0495-370. PMID 7585069
- [Result] Dotsch J, Demirakca S, Terbrack HG, Huls G, Rascher W, Kuhl PG. Airway nitric oxide in asthmatic children and patients with cystic fibrosis. Eur Respir J. 1996 Dec;9(12):2537-40. doi: 10.1183/09031936.96.09122537. PMID 8980966
- [Result] Ferguson EA, Eccles R. Changes in nasal nitric oxide concentration associated with symptoms of common cold and treatment with a topical nasal decongestant. Acta Otolaryngol. 1997 Jul;117(4):614-7. doi: 10.3109/00016489709113447. PMID 9288222
- [Result] Kharitonov SA, Rajakulasingam K, O'Connor B, Durham SR, Barnes PJ. Nasal nitric oxide is increased in patients with asthma and allergic rhinitis and may be modulated by nasal glucocorticoids. J Allergy Clin Immunol. 1997 Jan;99(1 Pt 1):58-64. doi: 10.1016/s0091-6749(97)70301-4. PMID 9003212
- [Result] Arnal JF, Didier A, Rami J, M'Rini C, Charlet JP, Serrano E, Besombes JP. Nasal nitric oxide is increased in allergic rhinitis. Clin Exp Allergy. 1997 Apr;27(4):358-62. PMID 9146927
- [Result] Lewis NS. Comparisons between mammalian and artificial olfaction based on arrays of carbon black-polymer composite vapor detectors. Acc Chem Res. 2004 Sep;37(9):663-72. doi: 10.1021/ar030120m. PMID 15379582
- [Result] Fens N, Zwinderman AH, van der Schee MP, de Nijs SB, Dijkers E, Roldaan AC, Cheung D, Bel EH, Sterk PJ. Exhaled breath profiling enables discrimination of chronic obstructive pulmonary disease and asthma. Am J Respir Crit Care Med. 2009 Dec 1;180(11):1076-82. doi: 10.1164/rccm.200906-0939OC. Epub 2009 Aug 27. PMID 19713445
- [Result] American Thoracic Society; European Respiratory Society. ATS/ERS recommendations for standardized procedures for the online and offline measurement of exhaled lower respiratory nitric oxide and nasal nitric oxide, 2005. Am J Respir Crit Care Med. 2005 Apr 15;171(8):912-30. doi: 10.1164/rccm.200406-710ST. No abstract available. PMID 15817806
- [Result] Clement PA, Gordts F; Standardisation Committee on Objective Assessment of the Nasal Airway, IRS, and ERS. Consensus report on acoustic rhinometry and rhinomanometry. Rhinology. 2005 Sep;43(3):169-79. PMID 16218509
- [Result] Serrano C, Valero A, Picado C. [Nasal nitric oxide]. Arch Bronconeumol. 2004 May;40(5):222-30. doi: 10.1016/s1579-2129(06)70088-x. No abstract available. Spanish. PMID 15117622